CLINICAL TRIAL: NCT02777450
Title: Validity and Predictive Value of Manual Clinical Test to Identify Symptomatic Segments in Lumbar Chronic Patients
Status: Completed | Type: Observational
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, santos caudevilla polo, Professor Unidad de Investigación de Fisioterapia, Universidad de Zaragoza
Other Study IDs: PI16/0015
Record Dates: First submitted 2016-05-05; First posted 2016-05-19 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Low Back Pain
Keywords: low back pain; physical examination; local anesthesia
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Block group: Lumbar facet block. Levobupivacaine 0,25% and corticosteroids
  Interventions: Procedure: lumbar facet block

INTERVENTIONS:
Procedure: lumbar facet block — injection of Levobupivacaine 0,25% and corticosteroids

SUMMARY:
This study evaluates the predictor value of manual test in lumbar chronic patients blocks. Bibliography has show limited evidence of clinical predictors in lumbar blocks. Prior to lumbar facet block or medial branch denervation patient will be evaluated with manual provocative segmental movements, lumbar sagittal range of motion, manual segmental movement and slump neural test . Immediate, one and six months effect will be registered.

DETAILED DESCRIPTION:
Clinical tests have sown limit evidence to predict efficacy of lumbar facet blocks. Segmental mobility tests have been included into the protocol to evaluate the efficacy of the lumbar blocks.

Chronic low back pain patients will be tested to evaluate the predictor value of manual clinical tests.

Patients from the "Lozano Blesa" Hospital pain clinic will be evaluate before, one month and six months after the lumbar facet block.

ELIGIBILITY:
Inclusion Criteria:

* more than 3 months of low back pain.
* lumbar with or without leg pain.
* patient treated with a lumbar facet block or medial nerve denervation.
* capable to be physically explored.
* capable to fill a questionaire.

Exclusion Criteria:

* no mechanical pain.
* severe medical condition.
* severe lumbar trauma.
* severe lumbar instability.
* severe lumbar deformity
* psychiatric disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic lumbar pain patients from the pain clinic service of the Lozano Blesa University Hospital
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Pain intensity Visual analogue scale | baseline before the block
Change of the Pain intensity one hour after the block | one hour after the block
Change of the pain intensity one month after the block | one month after the block
Change of the pain intensity six months after the block | six months after the block

SECONDARY OUTCOMES:
range of motion ROM | baseline before the block
  Measure of the pain free lumbar flexion and extension range of motion. Measured with single inclinometer in grades
Change of the range of motion ROM | one month after the block
  Measure of the pain free lumbar flexion and extension range of motion. Measured with single inclinometer in grades
Change of the range of motion ROM | six months after the block
  Measure of the pain free lumbar flexion and extension range of motion. Measured with single inclinometer in grades
lumbar segmental provocation manual test | baseline before the block
Change of the lumbar segmental provocation manual test | one month after the block
Change of the lumbar segmental provocation manual test | six months after the block
lumbar manual segmental joint play test | baseline before the block
Change of the lumbar manual segmental joint play test | one month after the block
Change of the lumbar manual segmental joint play test | six months after the block
Algometer: Pressure Pain threshold | baseline before the block
  Measure of the pressure pain threshold of the hand and the interspinous ligament from T12 to L5
Change of the Algometer: Pressure Pain threshold | one month after the block
  Measure of the pressure pain threshold of the hand and the interspinous ligament from T12 to L5
Change of the Algometer: Pressure Pain threshold | six months after the block
  Measure of the pressure pain threshold of the hand and the interspinous ligament from T12 to L5
oswestry disability index | baseline before the block
Change of the oswestry disability index | one month after the block
Change of the oswestry disability index | six months after the block
hospital anxiety and depression scale | baseline before the block
Change of the hospital anxiety and depression scale | one month after the block
Change of the hospital anxiety and depression scale | six months after the block
11 point global rating of change scale | one month after the block
Change of the 11 point global rating of change scale | 6 months after the block
Douleur Neuropathique 4 questionnaire | baseline before the block
Change of the Douleur Neuropathique 4 questionnaire | one month after the block
Change of the Douleur Neuropathique 4 questionnaire | six months after the block
slump neural test | baseline before the block
Change of the slump neural test | one month after the block
Change of the slump neural test | six months after the block

CONTACTS AND LOCATIONS:
Overall Officials: Elena Estébanez, Study Director — Universidad de Zaragoza
Locations (1):
- Universidad de Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No
Yes to the pain clinic service